CLINICAL TRIAL: NCT06594887
Title: Use of Rectal Spacers for Proton Beam Radiation Therapy for Localized Prostate Cancer: Prospective Clinical Study
Brief Title: Rectal Spacers Use in Prostate Cancer Radiation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Princeton ProCure management, LLC. (Other)
Responsible Party: Principal Investigator, Edward M. Soffen, M.D., Edward M. Soffen, M.D., Princeton ProCure management, LLC.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1378387
Record Dates: First submitted 2024-08-26; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SpaceOAR Vue (Experimental)
  Interventions: Device: SpaceOAR Vue
- BioProtect Balloon Implant System (Experimental)
  Interventions: Device: BioProtect Balloon Implant System

INTERVENTIONS:
Device: SpaceOAR Vue — Peri-rectal hydrogel spacer consists of a layer of polyethylene-glycol gel (SpaceOAR vue) in order to outdistance the prostate from anterior rectal wall
  Other Names: Hydrogel
  Arms: SpaceOAR Vue
Device: BioProtect Balloon Implant System — The balloon spacer is a biodegradable balloon made of poly (L-Lactide-co-caprolactone) which is a co-polymer of Poly Lactide acid and epsilon Caprolactone (BioProtect Balloon Implant System, BioProtect Ltd) inflated with saline, providing around 18 mm space height , and can be deflated and repositioned if needed, both laterally and along the distal /proximal planes, for optimal uniformity of spacing.
  Arms: BioProtect Balloon Implant System

SUMMARY:
This prospective, 2-arm clinical trial aims to evaluate the use of rectal spacers in patients with localized prostate cancer scheduled for Proton Beam Therapy (PBT). Up to 50 subjects will be enrolled in this study.

Study visits will include screening, spacer placement, treatment planning, end-of-treatment assessment, and follow-up visits at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria

1. Subjects greater than 18 years old with prostate cancer
2. Subjects must have histologically confirmed adenocarcinoma of the prostate with biopsy taken within 12 months and must be planned to undergo proton beam therapy with rectal spacer
3. Subjects must have clinical stage T1-T3 with no posterior extra capsular extension of the prostate cancer
4. PSA less than or equal to 20 ng/mL
5. Gleason Score less than or equal to 7
6. Capacity to comprehend and readiness to sign a written informed consent form

Exclusion Criteria

1. Planned Pelvic lymph node radiotherapy.
2. Metastatic disease.
3. Prior local prostate cancer therapy
4. Active Inflammatory bowel disease requiring treatment with steroids.
5. Prior radical prostatectomy.
6. Active urinary tract infection.
7. Acute or chronic inflammation or infection of the prostate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Perirectal distance | 2-4 months
  Perirectal distance evaluated by measurement of the prostate-rectum separation as measured on treatment planning CT simulation.

SECONDARY OUTCOMES:
Spacer stability over time | 2-4 months
  Evaluated by spacer's height (mm) measurements taken at the last radiation treatment day.
Mean rectal dose | 2-4 months
  Spacers effect on the exposure of the rectum to radiation (rV 70)

CONTACTS AND LOCATIONS:
Locations (1):
- Procure Proton Therapy Center, Somerset, New Jersey, United States